CLINICAL TRIAL: NCT05616442
Title: Ketotifen in Non-Alcoholic Fatty Liver Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Elberri, principal investigator and clinical professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E112022
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hepatic Disease
Keywords: Nonalcoholic fatty liver disease (NAFLD)
MeSH Terms: conditions — Digestive System Diseases; Non-alcoholic Fatty Liver Disease | interventions — Ketotifen; Vitamin E

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 as Vitamine E group (Experimental): Vitamin E as standard therapy
  Interventions: Drug: Vitamin E
- Group two as Ketotifen group (Experimental): Ketotifen as interventional
  Interventions: Drug: Ketotifen

INTERVENTIONS:
Drug: Ketotifen — Mast cell stabilizer
  Arms: Group two as Ketotifen group
Drug: Vitamin E — Dietary supplement
  Arms: Group 1 as Vitamine E group

SUMMARY:
The aim of this study is to investigate the safety and efficacy of using ketotifen in patients with NAFLD patients without cirrhosis

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is characterized by the accumulation and deposition of fats in the hepatocytes which affect the liver structure and function. Causes of NAFLD vary but mainly attributed to dyslipidemia and obesity. Prevalence of NAFLD has been raised over years from 25% in 2005 to over 37% in 2016 and continues to increase to become one of the most common chronic liver disease (Li J et al., 2019).

The disease progress from steatosis and inflammatory infiltration that is known as nonalcoholic steatohepatitis (NASH) to liver fibrosis, cirrhosis, and ultimately hepatocellular carcinoma. Despite these serious outcomes, no definitive known approved medication for NASH has been developed. NAFLD management is mainly dependent on diet control, physical activity, and some supportive treatments mainly to prevent the disease complications (Mundi et al., 2020).

Mast cells (MCs) are responsible releasing mediators, including preformed bioactive metabolites (histamine and tryptase,), newly synthesized cytokines [transforming growth factor beta (TGF-β), tumor necrosis factor alpha (TNF-α) (Pham et al., 2022). MCs can lead to microvesicular steatosis, ductal reaction (DR), biliary senescence, inflammation, angiogenesis, and liver fibrosis during NAFLD/NASH (Huang et al., 2022). Consequently, MC stabilizer such as ketotifen has emerged as promising approach to improve patients with NASH through its antioxidant and anti-inflammatory effects (Kim et al., 2014; Abdelzaher et al., 2020).

ELIGIBILITY:
-Inclusion criteria: Adult males or females aged ≥18 years.

* All patients are diagnosed to have fatty liver grading 1, 2 or 3 on abdominal ultrasound with Hepatic steatosis index > 36 to be considered as a NAFLD patient.
* Confirmed diagnosis of NASH
* Exclusion Criteria:
* Current or history of significant alcohol consumption.
* Use of drugs historically associated with nonalcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins).
* Prior or planned bariatric surgery.
* Uncontrolled diabetes defined as Hemoglobin A1c 9.5% or higher.
* Evidence of other forms of chronic liver disease as Hepatitis B, Hepatitis C, Wilson's disease, Alpha-1-antitrypsin (A1AT) deficiency, Hemochromatosis, drug-induced liver disease.
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial and breast feeding.
* Use of other drugs known to have possible positive effects on steatosis.
* Other anti-histaminic, sedating agents (CNS depressants) and anticholinergic medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
fibrosis improvement (≥ 1 stage) | up to 6 months
  F0: no fibrosis F1: portal fibrosis without septa by fibroscan

SECONDARY OUTCOMES:
improvement of inflammatory biochemical markers as TNF | up to 6 months
  tumor necrosis factor measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt